CLINICAL TRIAL: NCT01279473
Title: A Phase I/II Multicenter, Dose-escalation Study of Oral Nilotinib on a Continuous Daily Dosing Schedule in Adult Patients With Imatinib-resistant or Imatinib-intolerant Chronic Myelogenous Leukemia (CML), or Relapse/Refractory Ph+ALL (Philadelphia Positive Acute Lymphocytic Leukemia)(Extension Study)
Brief Title: Study to Evaluate Nilotinib in Adult Patients With Imatinib-resistant or Imatinib-intolerant Chronic Myelogenous Leukemia (CML), or Relapse/Refractory Ph+ Acute Lymphoblastic Leukemia (ALL) (Extension Study)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107A1101E1; TAS-3-01
Record Dates: First submitted 2010-12-02; First posted 2011-01-19 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2011-08

CONDITIONS: Chronic Myelogenous Leukemia; Acute Lymphoblastic Leukemia
Keywords: Chronic Myelogenous Leukemia; CML; Acute Lymphoblastic Leukemia; Philadelphia Chromosome Positive, ph+ ALL; Acute Lymphoblastic Leukemia (Philadelphia Chromosome Positive)
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — nilotinib

ARMS (1):
- Nilotinib (Experimental)
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib
  Other Names: AMN107

SUMMARY:
This study will investigate if nilotinib provides an improved safety and efficacy profile over that seen in patients receiving Imatinib.

ELIGIBILITY:
Inclusion Criteria:

* Patients who complete CAMN107A1101 and obtained Informed concent by document

Exclusion Criteria:

* None

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-08; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 3 weeks

SECONDARY OUTCOMES:
Best hematologic response rate and Best cytogenetic response rate. | 3 years
Percentage of BCR-ABL genes transcript and mutation status of BCR-ABL | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Aichi, Japan

REFERENCES:
- See also: Results from CAMN107A1101E1 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=4004